CLINICAL TRIAL: NCT00838656
Title: A Randomised Feasibility Study of Extended Chemotherapy With Neoadjuvant Carboplatin, Then Surgery Followed by Adjuvant Paclitaxel and Gemcitabine Verses Neoadjuvant Gemcitabine and Carboplatin, Then Surgery, Followed by Adjuvant Paclitaxel
Brief Title: Two Different Schedules of Carboplatin, Paclitaxel, Gemcitabine, and Surgery in Treating Patients With Newly Diagnosed Stage IIIC or Stage IV Primary Epithelial Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Warwick Medical School (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000632859; WMS-NEOESCAPE-AK/RH/22498/1; ISRCTN24742183; EUDRACT-2005-001875-37; EU-20904; MREC-07/Q2803/73; RG_05-003
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2011-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: ovarian carcinosarcoma; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Gemcitabine; Paclitaxel

ARMS (2):
- Arm I (Experimental): Patients receive carboplatin IV over 1 hour and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may undergo treatment with paclitaxel and may also receive 6 more courses of neoadjuvant chemotherapy. Patients may then undergo surgery. After surgery, patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel
- Arm II (Experimental): Patients receive carboplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may undergo treatment with paclitaxel and may also receive 6 more courses of neoadjuvant chemotherapy. Patients may then undergo surgery. After surgery, patients receive paclitaxel IV over 3 hours and gemcitabine hydrochloride IV over 30 minutes on day 1. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin — Given IV in one of two schedules
Drug: gemcitabine hydrochloride — Given IV in one of two schedules
Drug: paclitaxel — Given IV in one of two schedules

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, gemcitabine, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known which treatment regimen may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving one of two chemotherapy regimens containing carboplatin, gemcitabine, and paclitaxel works in treating patients undergoing surgery for newly diagnosed primary stage IIIC or stage IV ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine and compare the feasibility of two sequential neoadjuvant regimens in patients with newly diagnosed, stage IIIC-IV ovarian or peritoneal carcinoma.
* To confirm the feasibility of extended sequential regimens offering 6+6 courses of chemotherapy in patients presenting with inoperable disease.
* To establish the feasibility of biweekly paclitaxel with vs without gemcitabine hydrochloride in the adjuvant phase, after carboplatin neoadjuvant induction.

OUTLINE: This is a multicenter study. Patients are stratified according to serum albumin (< 30 g/dL vs 30-35 g/dL vs > 35 g/dL), FIGO stage (stage IIIC vs stage IV), and histological grade (well-differentiated [grade 1] vs moderately well-differentiated [grade 2] vs poorly differentiated [grade 3]). Patients are randomized to 1 of 2 treatment arms.

* Neoadjuvant therapy:

  * Arm I: Patients receive carboplatin IV over 1 hour and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive carboplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

In both arms, patients with disease progression are switched to adjuvant paclitaxel-based chemotherapy. Patients with responding disease after switching regimens may undergo debulking surgery at the investigator's discretion.

* Surgery: After completion of 6 courses of chemotherapy, all patients are evaluated for surgery. Patients with questionable operability based on clinical or radiological criteria are re-assessed laparoscopically. Patients judged to have disease that is amenable to optimal debulking at laparotomy are recommended for debulking surgery. Patients judged to have disease that is not amenable to optimal debulking are reconsidered for surgery after they receive an additional 6 courses of chemotherapy. Patients with disease progression after completion of 12 courses of chemotherapy undergo laparotomy only if there is a clinically pressing need to palliate their condition and if surgery offers some prospect of achieving this result (e.g., palliation for bowel obstruction).
* Adjuvant therapy:

  * Arm I: Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive paclitaxel IV over 3 hours and gemcitabine hydrochloride IV over 30 minutes on day 1. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete quality of life questionnaires at baseline, after completion of course 6 of neoadjuvant therapy, before course 7, and at the end of study treatment.

After completion of study therapy, patients are followed periodically for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically, radiologically, and histologically confirmed diagnosis of 1 of the following:

  * Primary epithelial ovarian cancer
  * Primary peritoneal carcinoma
  * Ovarian carcinosarcoma
  * Fallopian tube carcinoma
* Newly diagnosed, stage IIIC/IV disease with or without ascites
* None of the following histologies allowed:

  * Mucinous
  * Classic clear cell
  * Micropapillary or microacinar borderline tumors with or without invasive implants
* Unsuitable for primary debulking surgery, as defined by the following:

  * Laparoscopic or other minor surgical-staging procedures
  * Supplementary clinical and radiological assessments
* Presenting with factors affecting suitability for successful complete resection and necessarily prompting laparoscopic assessment, including any of the following:

  * CT scan or MRI evidence of peritoneal carcinomatosis, extensive mesenteric infiltration, diaphragmatic involvement, extensive retroperitoneal involvement, and cytologically verified malignant pleural effusion and/or ascites
  * Clinical evidence of ascites with radiological evidence of multisite disease
  * Clinical evidence of pelvic infiltration and radiological evidence of multisite disease
  * FIGO stage IV disease, including cervical/supraclavicular lymphadenopathy, intrahepatic parenchymal metastases, or cytologically confirmed malignant pleural effusion
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy ≥ 3 months
* WBC > 3.0/mm³
* Platelet count ≥ 100,000/mm³
* ANC ≥ 1,500/mm³
* AST and ALT < 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN
* Bilirubin < 1.5 times ULN
* Estimated glomerular filtration rate ≥ 30 mL/min
* No diabetics, hypertensive smokers, or other patients with pre-existing occult neuropathic deficits
* No poorly controlled, potentially serious medical conditions, including any of the following:

  * Cerebrovascular events within the past 12 months
  * Severe chronic respiratory conditions requiring prior hospitalization
  * Active infections
  * Poorly controlled seizures
  * Morbid psychiatric conditions likely to render treatment compliance with the protocol difficult
* No other malignancy treated with chemotherapy or radiotherapy except nonmelanoma skin cancer or carcinoma in situ of the cervix

  * Prior malignancies disease-free for > 5 years not treated with chemotherapy allowed
* No other reasons likely to cause inability to comply with treatment schedule and follow-up
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients completing 12 courses of chemotherapy

SECONDARY OUTCOMES:
Toxicity
Quality of life as assessed by FACT-G, FACT-0, and FACT-T periodically
Objective response rate to the neoadjuvant phase of chemotherapy (i.e., first 6 courses) as assessed by CT scan, by laparoscopy, clinically, and by CA-125 level
Objective response rate following all 12 courses of treatment assessed clinically, by CT scan, and by CA-125 level
Progression-free survival, particularly at 34 weeks
Overall survival, particularly at 34 weeks
Rates of optimal and suboptimal interval debulking

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Poole, MD, Principal Investigator — University Hospital Birmingham
Locations (4):
- United Kingdom (4):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Good Hope Hospital, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - New Cross Hospital, Wolverhampton, England